CLINICAL TRIAL: NCT01977170
Title: Phase 1 Study of Hib Vaccine (Bio Farma)
Brief Title: Safety of Hib Vaccine (Bio Farma)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Hib 0110
Record Dates: First submitted 2013-10-29; First posted 2013-11-06 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
Keywords: Adults; Hib vaccines; Immunogenicity; Safety
MeSH Terms: interventions — Haemophilus influenza type b polysaccharide vaccine-tetanus toxin conjugate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hib/PRP-T vaccine (Experimental): One dose, correspond to 0.5 ml, composed of:
  PRP-T 10ug NaCl 0.85%
  Frequency: 1 injection
  Interventions: Biological: Hib/PRP-T vaccine

INTERVENTIONS:
Biological: Hib/PRP-T vaccine — Hib liquid vaccine

SUMMARY:
The objective of this study was to know the safety of Hib/PRP-T vaccine and immediate reactions within the first 30 minutes after injection.

DETAILED DESCRIPTION:
This trial was an open-label study, no randomization, and no placebo or control group. Total 25 young healthy adult (volunteers) followed this trial. The safety was assessed within 24 hours, 48 hours, 72 hours, and 28 days after injection.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18 - 40 years old)
* Provision of written informed consent
* Good health according to the clinical investigator
* Willingness and ability to adhere to the regimen of the study

Exclusion Criteria:

* Known not enrolled in other study
* Pregnancy or lactation
* Known or suspected allergy to any of the vaccine component (by medical history)
* History of unusual reaction to any previous vaccination
* Known or suspected immune deficiency, or use of medication that may influence the immune system
* Prior respiratory infection
* Other vaccination during the study, or one week before (inactivated vaccine) or one month (live vaccine) before the study
* Acute febrile illness (temperature > 37.5 Celsius)
* Present evidence of serious diseases demanding medical treatment
* Any significant congenital or chronic disorder

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2010-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Incidence rate of adverse event of Hib vaccine (Bio Farma) | 30 minutes
  Local and systemic reactions

SECONDARY OUTCOMES:
To evaluate the antibody function serum using serum bactericidal activities test | 28 days
  Presence of serum of bactericidal activities after immunization.
Incidence rate of adverse event of Hib vaccine (Bio Farma) | 28 hours, 48 hours, 72 hours, 28 days
  Local and systemic reaction

CONTACTS AND LOCATIONS:
Overall Officials: Kusnandi Rusmil, PhD, Principal Investigator — Faculty of Medicine UNPAD
Locations (1):
- Hasan Sadikin Hospital, Bandung, West Java, Indonesia